CLINICAL TRIAL: NCT02912936
Title: A Medium Chain Triglyceride INTervention for Alzheimer Disease (A MINT for AD)
Brief Title: A Medium Chain Triglyceride Intervention for Patients With Alzheimer Disease
Acronym: MINT-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Haakon Nygaard, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H15-02537
Record Dates: First submitted 2016-07-13; First posted 2016-09-23 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer's Disease
Keywords: medium chain triglyceride; MCT; coconut oil; MRI; PET; ketones
MeSH Terms: conditions — Alzheimer Disease; Ketosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ketogenic medium chain triglyceride drink (Experimental): Lactose-free skim milk drink containing 25 g of MCT oil per 250 ml.
  Interventions: Dietary Supplement: Ketogenic medium chain triglyceride drink (MCT drink)
- Placebo (Placebo Comparator): Lactose-free skim milk drink containing high-oleic sunflower oil in the equivalent amount of energy as the active arm.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketogenic medium chain triglyceride drink (MCT drink) — 10 days supplementation with the MCT drink. Participants in dose group 1 will be assigned to 10 g per day, those in dose group 2 will be assigned 20 g per day, those in dose group 3 will be assigned 30 g per day, those in dose group 4 will be assigned 40 g per day, and those in dose group 5 will be assigned 50 g per day. The drink will be taken in the morning and evening. Participants will be enrolled 8 per group in ascending order.
  Arms: Ketogenic medium chain triglyceride drink
Dietary Supplement: Placebo — 10 days supplementation with the placebo drink. Participants in dose group 1 will be assigned to 10 g per day, those in dose group 2 will be assigned 20 g per day, those in dose group 3 will be assigned 30 g per day, those in dose group 4 will be assigned 40 g per day, and those in dose group 5 will be assigned 50 g per day. The drink will be taken in the morning and evening. Participants will be enrolled 8 per group in ascending order.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine safety, tolerability, and pharmacokinetics/dynamics of a ketogenic dietary supplement containing medium chain triglycerides (MCTs) in patients with Alzheimer disease (AD). Novel imaging and laboratory biomarkers in response to this intervention will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild-moderate Alzheimer disease (AD)
* Mini-Mental State Examination (MMSE) 16-26
* Study partner available who has frequent contact with the participant
* Good visual and auditory acuity for neuropsychological testing
* Education including completion of at least six grades
* Must read and speak English fluently
* Antidepressants permitted, if stable for 4 weeks prior to screening (and participant is not currently depressed and does not have a history of major depression within the past 1 year)
* Cholinesterase inhibitors permitted, if stable for 12 weeks prior to screening

Exclusion Criteria:

* Any significant neurologic disease other than AD
* History of Diabetes Mellitus type I or II
* Any contraindications to MRI or PET studies
* Major depression, bipolar disorder as described within the past 1 year.
* History of schizophrenia
* History of alcohol or substance abuse or dependence within the past 2 years
* Any significant systemic illness or unstable medical condition, which could lead to difficulty complying with the protocol
* Current use of specific psychoactive medications
* Investigational amyloid lowering therapies are prohibited two months prior to screening and for the duration of the trial. Other investigational agents are prohibited one month prior to screening and for the duration of the trial.
* History of brain cancer

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events, serious adverse events | From baseline to day 10 of intervention
Plasma ketone concentrations in response to ascending dose of MCT | Day 10 of intervention at 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, and 6 hours post MCT dose
  Plasma ketone concentrations of betahydroxybutyrate (BHB) and acetoacetate (AcAc) will be measured in response to MCT dosing from 10-50 grams daily.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of MCT | Day 10 of intervention at 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, and 6 hours post MCT dose
  To determine the MCT plasma concentration at stated time points in response to MCT dosing from 10-50 grams daily.

OTHER OUTCOMES:
Cerebral metabolic rate of glucose in response to a ketogenic MCT drink | Baseline and day 10 of intervention
  Assess changes in metabolic rate of glucose by 18F fludeoxyglucose positron emission tomography (FDG-PET) in response to escalating doses of MCT (10-50grams daily) in patients with Alzheimer's disease
Cerebral blood flow in response to a ketogenic MCT drink | Baseline and day 10 of intervention
  Assess changes in brain blood flow using MRI (Arterial Spin Labeling) in response to escalating doses of MCT (10-50 grams daily) in patients with Alzheimer's disease
Changes in MR Spectroscopy (N-acetylaspartate, glutamate, glutamine) in response to a ketogenic MCT drink | Baseline and day 10 of intervention
  Assess changes in brain chemistry (measuring (N-acetylaspartate, glutamate, glutamine) in response to MCT treatment across a dose range of 10-50grams daily
Changes in daily physical activity in response to a ketogenic MCT drink | Baseline and day 10 of intervention
  Changes in behavior rhythms (activity level and sleep/rest) in response to MCT treatment across a dose range of 10-50grams daily, using an actigraphy watch.

CONTACTS AND LOCATIONS:
Overall Officials: Haakon Nygaard, MD, PhD, Principal Investigator — University of British Columbia; Howard Feldman, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia, Canada